CLINICAL TRIAL: NCT00556595
Title: Circumferential Pulmonary Vein Ablation in Paroxysmal Atrial Fibrillation: Randomized Comparison Between a Primary Anatomical Versus a Primary Electrophysiological Approach
Brief Title: Primary Anatomical Versus Primary Electrophysiological Approach in Circumferential Pulmonary Vein Ablation
Acronym: CPVA-PAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bonn (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPVA-PAF; IRB 160/07
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: atrial fibrillation; paroxysmal; symptomatic; drug-refractory
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): primary electrophysiological approach
  Interventions: Procedure: primary electrophysiological approach
- 2 (Active Comparator): primary anatomical approach
  Interventions: Procedure: primary anatomical approach

INTERVENTIONS:
Procedure: primary electrophysiological approach — primary ablation of atrio-venous breakthrough sites followed by circumferential ablation around pulmonary vein orifice
  Arms: 1
Procedure: primary anatomical approach — primary circumferential ablation around the pulmonary vein orifice followed by ablation of possible conduction gaps
  Arms: 2

SUMMARY:
Randomized comparison between 2 techniques of circumferential pulmonary vein ablation in paroxysmal atrial fibrillation: Primary anatomical ablation with secondary closure of possible electrical gaps versus primary electrophysiological ablation at the sites of atrio-venous electrical breakthroughs with secondary circumferential ablation around the pulmonary vein orifice

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal atrial fibrillation
* age over 18 years

Exclusion Criteria:

* persistent atrial fibrillation
* reversible cause of atrial fibrillation
* inability to comply with follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-11; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial tachyarrhythmias at 6-months follow-up | 6 months

SECONDARY OUTCOMES:
Comparison of procedural characteristics (duration, fluoroscopy time, ablation time, ablation energy, complications) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lars M Lickfett, MD, Principal Investigator — University Hospital Bonn, Department of Cardiology

REFERENCES:
- [Background] Oral H, Scharf C, Chugh A, Hall B, Cheung P, Good E, Veerareddy S, Pelosi F Jr, Morady F. Catheter ablation for paroxysmal atrial fibrillation: segmental pulmonary vein ostial ablation versus left atrial ablation. Circulation. 2003 Nov 11;108(19):2355-60. doi: 10.1161/01.CIR.0000095796.45180.88. Epub 2003 Oct 13. PMID 14557355
- [Background] Arentz T, Weber R, Burkle G, Herrera C, Blum T, Stockinger J, Minners J, Neumann FJ, Kalusche D. Small or large isolation areas around the pulmonary veins for the treatment of atrial fibrillation? Results from a prospective randomized study. Circulation. 2007 Jun 19;115(24):3057-63. doi: 10.1161/CIRCULATIONAHA.107.690578. Epub 2007 Jun 11. PMID 17562956
- [Background] Karch MR, Zrenner B, Deisenhofer I, Schreieck J, Ndrepepa G, Dong J, Lamprecht K, Barthel P, Luciani E, Schomig A, Schmitt C. Freedom from atrial tachyarrhythmias after catheter ablation of atrial fibrillation: a randomized comparison between 2 current ablation strategies. Circulation. 2005 Jun 7;111(22):2875-80. doi: 10.1161/CIRCULATIONAHA.104.491530. Epub 2005 May 31. PMID 15927974